CLINICAL TRIAL: NCT03846778
Title: Risk Factors of Complications After Ileocolic Resection for Crohn Disease According to the Comprehensive Complication Index - RICCI
Brief Title: Risk Factors of Complications After Ileocolic Resection for Crohn Disease According to the Comprehensive Complication Index
Acronym: RICCI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0050
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Crohn Disease; Ileocolic Resection
Keywords: Postoperative outcomes; Laparoscopy; Comprehensive complication index; Postoperative complications
MeSH Terms: conditions — Crohn Disease; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Cytolyt Samples:
  Liquid conservation samples from patients who underwent endoscopic ultrasound with fine needle aspiration/biopsy for suspicious pancreatic mass at the CHU de Montpellier were conserved at +4°c.
  Cytolyt samples do not contain any cell or tissue from patient, this liquid is systematically trashed in current practice. No genetics analysis will be performed from these particular samples in the present study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim: The aim of this study was to investigate the risks factors of complications after ileocolic resection for Crohn disease according to the comprenhensive complication index.

Methods: Data collected between January 2010 and March 2020 will be analyzed. Informations about preoperative, peroperative and post operative will be collected. The outcome after surgery will be analysed according to the comprehensive complication index.

DETAILED DESCRIPTION:
There are several risk factors reported for postoperative complication after ileocolic resection for Crohn disease. With recent new therapeutics (anti TNF, monoclonal antibodies), these criteria are questioned.

According to the ECCO 2010 Consensus Conference, five post-operative risk factors for recurrence of Crohn disease were described: smoking, extensive small bowel resection (> 50cm), repeat bowel resection, presence of ano-perineal lesions, and penetrating disease (type B3). However, postoperative complication risk factors after ileocolic resection remain debated. Currently the place of a pre-operative treatment with anti-TNF seems to be a post-operative complication risk factor according to the last ECCO 2017 consensus conference, as well as preoperative parenteral nutrition and emergency versus planned surgery. In addition, a recent GETAID study seems to challenge the penetrating phenotype as a risk factor of postoperative complication. A current study could provide new data on the various known or suspected complication risk factors in the anti-TNF/monoclonal antibodies era.

The classification of Clavien Dindo does not necessarily take into account the respective severities of each complication in a patients. The new classification (Comprehensive Complication Index (CCI)) could be usefull to take into account all the complications and their importance, without focusing only on the most important. To our knowledge, there is no study specifically evaluating CCI after ileocolic resection for Crohn disease. We believe that the CCI can provide a more refined analysis of risk factors for postoperative complications after this procedure.

The aim of this study is to analyze the different complication risk factors after ileocecal resection according to the recent Comprehensive Complication Index, tools potentially more sensitive than Clavien Dindo classification to highlight differences in postoperative morbidity.

ELIGIBILITY:
Inclusion criteria:

* Patients who underwent an ileocolic resection for Crohn disease
* Patient ≥18 years old

Exclusion Criteria:

- Patient who reject the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring an ileocolic resection for Crohn disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 90 days (after surgery)
  Comprehensive Complication Index (CCI)

SECONDARY OUTCOMES:
Morbidity according to the Clavien Dindo Classification | 90 days (after surgery)
  Morbidity according to the Clavien Dindo Classification
Mortality | 90 days (after surgery)
  Mortality
Reoperation rate | 90 days (after surgery)
  Reoperation rate
Readmission rate | 90 days (after surgery)
  Readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France